CLINICAL TRIAL: NCT02219113
Title: Effectiveness and Safety of Intraarticular Administration of Autologous Adipose-Derived Regenerative Cells for Treatment of Degenerative Damage of Knee Articular Cartilage
Brief Title: Effectiveness and Safety of Autologous ADRC for Treatment of Degenerative Damage of Knee Articular Cartilage
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Central Clinical Hospital w/Outpatient Health Center of Business Administration for the President of Russian Federation (Other Government)
Collaborators: I.M. Sechenov First Moscow State Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RU-CCH-03-02-14
Record Dates: First submitted 2014-08-15; First posted 2014-08-18 (Estimated); Last update posted 2017-07-21 (Actual); Status verified 2017-07

CONDITIONS: Knee Joint Osteoarthritis
Keywords: Damage of articular cartilage; Cartilage degeneration; Intraarticular injection; ADRC; Adipose-derived regenerative cells; Adipose tissue; Stem cells
MeSH Terms: interventions — Arthroscopy; Lipectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ADRC injection (Experimental): Subjects will undergo liposuction under local anesthesia. Lipoaspirate will be processed to isolate and concentrate adipose-derived regenerative cells (ADRC). After ADRC isolation autologous cells suspension will be injected intraarticularly into knee joint.
  Interventions: Procedure: Arthroscopic surgery; Procedure: Liposuction; Device: ADRC isolation; Other: Intraarticular administration of autologous ADRC

INTERVENTIONS:
Procedure: Arthroscopic surgery
Procedure: Liposuction
Device: ADRC isolation — ADRC isolation performed using Celution 800/CRS System (Cytori Therapeutics Inc) according to manufacturer's protocol
Other: Intraarticular administration of autologous ADRC

SUMMARY:
Autologous adipose-derived regenerative cells (ADRC) extracted using Celution 800/CRS System (Cytori Therapeutics Inc) from a portion of the fat harvested from the patient's front abdominal wall. ADRC will be administered one-time intraarticularly. This is a single arm study with no control. All patients receive cell therapy.

DETAILED DESCRIPTION:
Patients with verified diagnosis knee joint osteoarthritis (degenerative damage of knee articular cartilage) will undergo knee arthroscopic debridement. 28 days later patients will will undergo liposuction from front abdominal wall under local anesthesia. After that autologous ADRC will be extracted using Celution 800/CRS System (Cytori Therapeutics Inc) from harvested adipose tissue. Extracted ADRC will be administered one-time intraarticularly.

ELIGIBILITY:
Inclusion Criteria:

* Pain in the knee joint during more than a half day assessed by VAS (score more than 40 mm)
* At least three of the following 6 criteria: 50 years of age or older, stiffness lasting less than 30 minutes, crepitus, bony tenderness, bony enlargement, no warmth to the touch
* Patient is able to walk without assistance
* Patient is familiar with Participant information sheet
* Patient signed informed consent form

Non-inclusion Criteria:

* Medical history of endoprosthetic knee replacement
* Medical history of lower extremity osteotomy
* Medical history of knee surgery (including arthroscopy) during preceding 1 year prior to enrollment
* Medical history of intraarticular injections during preceding 6 months prior to enrollment
* Secondary osteoarthritis of the knee joint: posttraumatic osteoarthritis (developed after clinically significant injury), intra-articular fractures, clinically significant varus or valgus deformities of lower limbs, septic arthritis, joint's inflammatory disorders, gout, advanced chondrocalcinosis, Paget's disease, ochronosis, acromegaly, hemochromatosis, Wilson's disease, primary synovial osteochondromatosis, osteonecrosis, hemophilia
* Patients prescribed for immunosuppressive treatment
* Medical history of systemic autoimmune and inflammatory diseases
* Significant weight loss (> 10% of body weight in the previous year) of unknown etiology
* Medical history of venous thromboembolism or estimated high risk of venous thromboembolism
* Patients prescribed for systemic corticosteroids or other medications treatment with proven impact on bone or cartilage tissue metabolism
* Clinically significant abnormalities in results of laboratory tests
* Any conditions limiting compliance (dementia, neuropsychiatric disease, drug and alcohol abuse etc.)
* Participation in other clinical trials (or administration of investigational drugs) during 3 months prior inclusion
* Patients with malignant tumors including postoperative period, patients receiving chemotherapy and/or radiotherapy.
* Patient's activated partial thromboplastin time exceeds normal levels more than 1,8 times
* Patients prescribed for anticoagulants treatment or patient received anticoagulants at least one hour prior lipoaspiration
* Medical history of heterotopic ossifications
* Patients prescribed for glycoprotein inhibitors treatment

Exclusion Criteria:

* Patient's refusal from the further participation in trial
* Patient's refusal from compliance with the requirements of contraception during the participation in research
* Chronic kidney disease IV- V stages (creatinine clearance < 30 mL/min estimated by Cockroft-Gault formula)
* Confirmed syphilis, HIV, hepatitis B or C infections

Dropout Criteria:

* Pregnancy

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2014-07; Primary Completion 2016-12 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Number of serious adverse events (SAEs) and serious adverse reactions (SARs) | 4 weeks after treatment
  Types, probability and severity of treatment emergent serious adverse events (SAEs) and serious adverse reactions (SARs)

SECONDARY OUTCOMES:
Quality of life monitoring | Follow up to completion (up to 24 weeks after treatment)
  Quality of life estimated by validated questionnaires: the Short Form (36) Health Survey (SF-36), Knee Injury and Osteoarthritis Outcome Score (KOOS)
Knee pain intensity monitoring | Follow up to completion (up to 24 weeks after treatment)
  Knee pain intensity assessed by Visual Analogue Scale (no pain=0; maximum pain=100 mm)
Changes in knee joint structures | Follow up to completion (up to 24 weeks after treatment)
  Changes in knee joint structure assessed by:
  1. X-ray (joint space width, bone contour, presence of osteophytes and sclerosis);
  2. MRI (articular cartilage, osteophytes, bone marrow abnormality, meniscal integrity, synovial effusion/tissue, anterior and posterior cruciate ligaments, and medial and lateral collateral ligaments);
  3. Ultrasonography (effusion, synovial thickening or hypertrophy, cartilage parameters, vascularity, Baker's cysts, osteophytes, tendon and ligament abnormalities, meniscal changes, bursitis, erosions and panniculitis)
Changes in knee function | Follow up to completion (up to 24 weeks after treatment)
  Changes in knee function assessed by validated questionnaire: Knee Society Score (KSS)

CONTACTS AND LOCATIONS:
Overall Officials: Sergey V Ivannikov, Professor, Principal Investigator — I.M. Sechenov First Moscow State Medical University; Ilya I Eremin, MD, PhD, Principal Investigator — Federal State Budgetary Institution "Central Clinical Hospital with Outpatient Health Center" of the Business Administration for the President of the Russian Federation; Center for Biomedical Technologies
Locations (1):
- Federal State Budgetary Institution "Central Clinical Hospital with Outpatient Health Center" of the Business Administration for the President of the Russian Federation; Center for Biomedical Technologies, Moscow, Russia